CLINICAL TRIAL: NCT02759003
Title: Nightime Noninvasive Mechanical Ventilation Initiation in Amyotrophic Lateral Sclerosis in an Outpatient Setting. A Non-inferiority Study.
Brief Title: Nightime NIV Initiation in Amyotrophic Lateral Sclerosis in an Outpatient Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Salvatore Maugeri (Other)
Collaborators: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Enrica Bertella, Principal Investigator, Fondazione Salvatore Maugeri
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTS 02/2011
Record Dates: First submitted 2016-04-27; First posted 2016-05-03 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-04

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- inpatients group (Active Comparator): In-hospital nightime NIV initiation. For the inpatients Group, NIV was initiated in the respiratory wards of the two hospitals and continued during night for a minimum of 4 hours/night.
  Inpatients had a 24-h availability of health staff care. During the night, they had nurses and physicians available on-hand.
  Interventions: Procedure: Nightime NIV initiation
- outpatients group (Experimental): Home nightime NIV initiation. For the outpatients group, diurnal NIV was initiated during a scheduled visit in a hospital dedicated room(at least 4 hours/day of care), the trial proceeded at home during the night with a personal caregiver.
  A minimum of 4 hours/night was required. No support during the night was provided to these patients.
  Interventions: Procedure: Nightime NIV initiation

INTERVENTIONS:
Procedure: Nightime NIV initiation — In-hospital vs home

SUMMARY:
In patients with amyotrophic lateral sclerosis (ALS), non-invasive mechanical ventilation (NIV) is usually initiated in an in-hospital regime. The investigators evaluated if NIV initiated in an outpatient setting can be as effective as regards patients' adherence. The investigators also evaluated factors predicting NIV adherence and disease progression.

DETAILED DESCRIPTION:
All patients with a definite ALS diagnosis, aged > 18 years, referred to the ALS outpatient clinics of the Fondazione Salvatore Maugeri Institute of Lumezzane (Brescia) and Istituto Don Gnocchi Onlus (Milano), Italy, for respiratory functional assessments for the purpose of early initiation of NIV were considered. Patients who were in clinically stable condition and without chest infections during the previous 3 months were considered eligible for the study.

Between March 2011 and March 2014, during an outpatient visit, the patients were randomized 1:1 to two groups for NIV initiation: outpatient vs. inpatient protocol.

In both groups a diurnal NIV initiation trial was performed using pressure-support ventilators in spontaneous/timed mode with a preset tidal volume (300 ml/kg) and a fixed back-up respiratory rate (12 breaths/min). The trial included: choice of the mask, setting of ventilator pressure, at least 2 hours of NIV under supervision.

Then, the patients underwent the nighttime NIV initiation trial for a maximum of 20 nights according to the outpatient vs. inpatient protocol.

NIV trial was stopped when: 1) patients used NIV > 4 hours/night for 3 consecutive nights, 2) patients and caregivers were able to manage with ventilator, 3) patients failed after 10 consecutive educational sessions.

At enrollment (T0), the end of NIV initiation trial (T1) and after 3 months from the end of the trial (T2) respiratory function tests, blood gas analysis, and sleep study were performed.

At T1 the investigators assessed NIV acceptance (as a minimum of 3 consecutive days >4 h/night), and dyspnea symptoms by VAS (day/night), staff and patients' satisfaction.

At T2: NIV adherence (>120 h/month) and patients' satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients
* definite ALS diagnosis
* aged > 18 years
* in clinically stable condition
* referred to the ALS outpatient clinics of the Fondazione Salvatore Maugeri Institute of Lumezzane (Brescia) and the Istituto Don Gnocchi Onlus (Milano), Italy for respiratory functional assessment for the purpose of early initiation of NIV
* no chest infections during the previous 3 months.

Exclusion Criteria:

* cognitive impairment
* refusal to participate
* severe comorbidities and contraindications to NIV (arrhythmias, cardiac failure, history of pneumothorax)
* distance from hospital > 40 km, travel problems to attend the outpatient clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-03; Primary Completion 2013-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Adherence as measured by the use of ventilator (hours/month) | At 3 months
  Evaluation after 3 months from the end of NIV initiation trial (T2)

SECONDARY OUTCOMES:
Changes in respiratory function as assessed by spirometry | At 3 months
  Evaluation at 3 months from the end of NIV initiation trial (T2)
Changes in dyspnea symptoms as assessed by Visual Analogue Scale | At 3 months
  Evaluation at 3 months from the end of NIV initiation trial (T2)
Patient's questionnaire of satisfaction | At 20 days
  Evaluation at the end of NIV initiation trial (T1)
Changes in respiratory function as assessed by Maximal inspiratory pressure/Maximal expiratory pressure | At 3 months
  Evaluation at 3 months from the end of NIV initiation trial (T2)
Changes in respiratory function as assessed by blood gas analysis | At 3 months
  Evaluation at 3 months from the end of NIV initiation trial (T2)

CONTACTS AND LOCATIONS:
Overall Officials: Enrica Bertella, MD, Principal Investigator — Fondazione Salvatore Maugeri

IPD SHARING:
Plan to Share IPD: No